CLINICAL TRIAL: NCT05871671
Title: The Effects of Pulmonary Rehabilitation on Bone Mineral Density in Patients Diagnosed With Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malta (Other)
Responsible Party: Principal Investigator, Melanie Axiak, Principal Investigator, University of Malta
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of Malta
Record Dates: First submitted 2023-05-13; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary Rehabilitation, Exercise, Physical Activity, Chronic Obstructive Pulmonary Disease, Osteoporosis, Bone Mineral Density and Bone Mineral Status
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Osteoporosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The control group shall consist of a minimum of 40 patients with a confirmed diagnosis of COPD and osteoporosis or osteopenia. This group which shall consist of patients who do not wish to participate in Pulmonary Rehabilitation but show the wish to form part of this study, or participants who are on the waiting list to be enrolled into the Rehabilitation classes, shall act as a control for the study and therefore not undergo PR and the following maintenance home exercise programme until completion of the study. All patients were medically stable and referred by their caring respiratory consultant.
  Interventions: Other: Control
- Active group (Experimental): The active group shall consist of a minimum of 40 patients with a confirmed diagnosis of COPD and osteoporosis or osteopenia. All patients shall receive a 16-week twice weekly PR programme which shall be followed by a 36-week maintenance home exercise programme. All patients were medically stable and referred by their caring respiratory consultant.
  Interventions: Behavioral: Pulmonary Rehabilitation

INTERVENTIONS:
Behavioral: Pulmonary Rehabilitation — A 16-week PR programme shall be delivered twice weekly to the active group. This shall be followed by a 36-week maintenance home exercise programme which shall be monitored every 4 weeks via a phone call from the researcher herself for 36 weeks. The subjects shall self-document their adherence to the home exercise programme on a diary which shall be returned to the researcher at week 52.
  Other Names: Respiratory Rehabilitation
  Arms: Active group
Other: Control — The control group shall not receive the 16-week PR programme and the following 36-week maintenance home exercise programme until completion of the study.
  Arms: Control group

SUMMARY:
Exercise has been reported to lead to improvements in Bone Mineral Density (BMD), however studies looking into the effects of exercise on BMD in Chronic Obstructive Pulmonary Disease (COPD) patients are still very limited. In view of this, the aims of such a study are to identify whether a 16-week Pulmonary Rehabilitation programme leads to improvements in BMD in patients with osteopenia and osteoporosis diagnosed with stable COPD, something which is warranted to reduce the risk of fractures and their related adverse consequences in these patients.

DETAILED DESCRIPTION:
Patients suffering from Chronic Obstructive Pulmonary Disease (COPD) are reported to have a high prevalence rate and increased risk of osteopenia and osteoporosis especially due to the intake of corticosteroids, a factor which increases their risks of falls and likelihood of fractures. Considering the enormous impact of such fractures on COPD patients, prophylactic measures are warranted to prevent further loss of BMD to reduce their risk of fractures and their related adverse consequences. Exercise has been reported to lead to improvements in BMD. Evidence regarding the effects of such an intervention on BMD in COPD patients is still very limited. In view of this, the aims of such a study are to identify whether a 16-week Pulmonary Rehabilitation (PR) programme leads to improvements in BMD in patients with osteopenia and osteoporosis diagnosed with stable COPD.

A minimum of 80 patients shall be allocated to either the active group or the control group by the intermediary. The active group shall receive a PR Programme delivered twice weekly for a period of 16 weeks which shall be followed by a maintenance home exercise programme for a period of 36 weeks. The other group which shall consist of patients who do not wish to participate in Pulmonary Rehabilitation but show the wish to form part of this study, or participants who are on the waiting list to be enrolled into the Rehabilitation classes, shall act as a control for the study and therefore not undergo PR and the following maintenance home exercise programme until completion of the study.

As part of the assessment, at baseline (week 0), demographic and anthropometric details and individual patient factors known to affect bone metabolism including; age, gender, smoking status and any concurrent prescribed medications and supplements, shall be gathered directly from all participants. The patients' body weight and height and the Body Mass Index shall be then calculated. Each participant's last DEXA scan measurement shall be retrieved from the Picture Archiving and Communication System (PACS) through the intermediary. All participants shall also have their functional mobility level and fall risk assessed using the Timed "Up and Go" test (TUGT). Estimated 10-year probability of hip fractures and major osteoporotic fractures shall be predicted using WHO web-based fracture risk assessment (FRAX) tool. All participants shall also have their functional exercise capacity assessed using the Six-Minute Walk Test (6MWT).

At week 16 and at week 52 all patients shall be reassessed as baseline, except for the measurement of the bone mineral density which shall be taken using DEXA scan only at week 52 and shall be retrieved from the PACS through the intermediary for the active and control group subjects and shall be required per protocol.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COPD by Spirometry
* Stable COPD confirmed by lack of an exacerbation within the 3 months preceeding the start of the study
* Confirmed diagnosis of osteopenia or osteoporosis by DEXA scan which would have been carried out at some point in the previous 12 months
* Due for a DEXA scan in the timeframe when the researcher shall be carrying out her data collection. This will ensure that no patients shall be receiving any exposures that were not part of their routine medical management
* Optimal medical management
* SpO2 >92% at rest
* Motivated and committed
* Suitable cognitive and communicative ability

Exclusion Criteria:

* Acute infection or exacerbation within the 3 months preceeding the start of the study
* Lack of motivation and non-adherence
* Unstable cardiovascular system

  * Myocardial Infarction within last 6 weeks
  * Uncontrolled hypertension
  * Unstable angina
  * Aortic stenosis
  * Acute Left Ventricular Failure
  * Uncontrolled cardiac arrhythmias
* Unstable diabetes
* Uncontrolled rheumatoid arthritis
* Severe orthopaedic or neuromuscular conditions
* Significant cognitive or psychiatric impairment which interfere with the PR programme

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The Changes in BMD | Change in BMD scores from baseline to 52weeks
  BMD scores measured by DEXA Scan

SECONDARY OUTCOMES:
Timed "Up and Go" Test (TUGT) | Change in TUGT scores from baseline to 16 weeks and from 16weeks to 52weeks
  A test to measure the functional mobility level and risk for falls
The fracture risk assessment (FRAX) tool | Change in FRAX tool scores from baseline to 16 weeks and from 16weeks to 52weeks
  A tool to estimate 10-year probability of hip fractures and major osteoporotic fractures
6 minute walk test (6MWT) | Change in 6MWT scores from baseline to 16 weeks and from 16weeks to 52weeks
  A walk test to assess the functional exercise capacity
Demographics, Anthropometrics and Medical Data | Change in Demographics, Anthropometrics and Medical Data from baseline to 16weeks and from 16weeks to 52weeks
  demographic and anthropometric details and individual patient factors known to affect bone metabolism including; age, gender, smoking status and any concurrent prescribed medications and supplements, shall be gathered directly from all participants. The patients' body weight and height and the Body Mass Index shall be then calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Axiak, BSc, Principal Investigator — University of Malta